CLINICAL TRIAL: NCT06575959
Title: An Open-Label, Single-Dose Clinical Study to Evaluate the Pharmacokinetics of Enlicitide in Participants With Hepatic Impairment
Brief Title: A Clinical Study of Enlicitide Decanoate in People With Liver Function Problems (MK-0616-030)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0616-030; MK-0616-030 (Other: MSD)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Insufficiency; Hepatic Impairment
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (HI) (Experimental): Participants will receive a single oral dose of enlicitide on Day 1
  Interventions: Drug: Enlicitide
- Healthy Controls (Experimental): Participants will receive a single oral dose of enlicitide on Day 1
  Interventions: Drug: Enlicitide
- Mild HI (Experimental): Participants will receive a single oral dose of enlicitide on Day 1
  Interventions: Drug: Enlicitide

INTERVENTIONS:
Drug: Enlicitide — Oral tablet
  Other Names: enlicitide decanoate; MK-0616/sodium caprate

SUMMARY:
Researchers have designed a new study medicine called enlicitide decanoate as a new way to lower the amount of low-density lipoprotein cholesterol (LDL-C) in a person's blood. Enlicitide decanoate will be called "enlicitide" from this point forward,

The purpose of this study is to learn what happens to enlicitide in a person's body over time (a pharmacokinetic or PK study). Researchers will compare what happens to enlicitide in the body when it is given to people with hepatic impairment (HI- meaning the liver does not work properly) and people who are in good health.

This study will have 2 parts. In Part 1, enlicitide will be given to people with moderate HI and people who are in good health. After Part 1, researchers may decide to include people who have mild HI and compare what happens to enlicitide in the body with people who are in good health.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

All participants:

* Has been a non-smoker or moderate smoker (≤ 10 cigarettes per day or equivalent) for at least 3 months prior to starting the study
* Has body mass index (BMI) ≥ 18.0 and ≤ 40.0 kg/m2

Participants with moderate or mild HI:

* Diagnosis of chronic (> 6 months) and stable (no sudden or severe episodes of illness due to worsening liver function in the past 2 months) hepatic insufficiency, and features cirrhosis (liver scarring) due to any cause.
* Is generally in good health with the exception of HI.

Healthy Control Participants:

* Medically healthy with no clinically significant medical history, physical examination, or clinical laboratory profiles

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

All participants:

* History of gastrointestinal disease which may affect food and drug absorption, or has had a gastric bypass or similar surgery.
* History of cancer
* Consumes greater than 3 servings of alcoholic beverages per day.
* Is on statin background therapy.

Participants with moderate or mild HI:

* Severe complications of liver disease within 3 months of entering the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Part 1: Area under the concentration versus time curve from 0 to infinity (AUC0-inf)AUC0-inf of enlicitide | Pre-dose and at designated time points up to 168 hours post dose
  AUC0-inf of enlicitide in plasma will be determined.
Part 1: Maximum concentration (Cmax) of enlicitide | Predose, and at designated timepoints up to 168 hours post-dose
  Cmax of enlicitide in plasma will be determined
Part 2: AUC 0-inf of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  AUC 0-inf of enlicitide in plasma will be determined
Part 2: Cmax of enlicitide | Predose, and at designated timepoints up to 168 hours post-dose
  Cmax of enlicitide in plasma will be determined

SECONDARY OUTCOMES:
Part 1: Area under the concentration versus time curve from 0 to 24 hours (AUC0-24) of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  AUC0-24 of enlicitide in plasma will be determined.
Part 1: Area under the concentration versus time curve from 0 to the time of the last quantifiable sample (AUC0-last) of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  AUC0-last of enlicitide in plasma will be determined
Part 1: Time to maximum (Tmax) observed plasma drug concentration of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  Tmax of enlicitide in plasma will be determined
Part 1: Apparent terminal half-life (t1/2) of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  t1/2 of enlicitide in plasma will be determined
Part 1: Apparent clearance (CL/F) of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  CL/F of enlicitide in plasma will be determined
Part 1: Apparent volume of distribution during terminal phase (Vz/F) of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  Vz/F of enlicitide in plasma will be determined
Part 1: Number of participants who experience one or more adverse events (AEs) | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 1: Number of participants who discontinue study intervention due to an AE | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 2: AUC0-24 of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  AUC0-24 of enlicitide in plasma will be determined.
Part 2: AUC0-last of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  AUC0-last of enlicitide in plasma will be determined
Part 2: Tmax observed plasma drug concentration of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  Tmax of enlicitide in plasma will be determined
Part 2: t1/2 of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  t1/2 of enlicitide in plasma will be determined
Part 2: CL/F of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  CL/F of enlicitide in plasma will be determined
Part 2: Vz/F of enlicitide | Pre-dose and at designated timepoints up to 168 hours post dose
  Vz/F of enlicitide in plasma will be determined
Part 2 Number of participants who experience one or more adverse events (AEs) | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Part 2: Number of participants who discontinue study intervention due to an AE | Up to approximately 6 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida
  - The Texas Liver Institute ( Site 0001), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com